CLINICAL TRIAL: NCT00397670
Title: A Multicenter Open-Label Study of the Safety and Contraceptive Efficacy of BufferGel® Spermicide Used With Diaphragm
Brief Title: Open Label Study of the Safety and Contraceptive Efficacy of BufferGel® With Diaphragm
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ReProtect Inc (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Premier Research (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCN 003OL
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2006-11-09 (Estimated); Status verified 2006-11

CONDITIONS: Contraception
MeSH Terms: interventions — BufferGel; Contraceptive Devices, Female

INTERVENTIONS:
Drug: Drug: BufferGel® with diaphragm

SUMMARY:
The purpose of this study is to study the safety and contraceptive effectiveness of BufferGel used with a contraceptive diaphragm.

ELIGIBILITY:
Inclusion Criteria:

* be healthy women, who are sexually active, at risk for pregnancy and desiring contraception
* be within the age range of 18 through 40 years inclusive
* be at low-risk for human immunodeficiency virus (HIV) or sexually transmitted disease (STD) infection, currently have (≥4 months) a single sexual partner who is also at low-risk for HIV or STD infection and expect to have the same partner for the duration of the study
* have a negative urine pregnancy test at the admission visit
* have normal cyclic menses with a usual length of 24 to 35 days over the last 2 months
* have a documented history of at least one spontaneous, normal menstrual cycle (two menses) since delivery, abortion, or after discontinuing hormonal contraception/hormonal therapy
* be willing to accept a risk of pregnancy
* be willing to engage in at least 4 acts of heterosexual vaginal intercourse per cycle for a period of approximately seven months
* be willing to be randomized to either study treatment as applicable
* be willing to be fitted with a diaphragm and use the diaphragm with test product during all acts of heterosexual vaginal intercourse for the duration of the study
* be willing to only use the test product with diaphragm as the primary method of contraception over the course of the study [with the exception of emergency contraception pills (ECPs), when indicated]
* be capable of using the product and diaphragm properly and agree to observe all study directions and requirements

Exclusion Criteria:

* have a history of allergy or sensitivity to spermicides, products containing N-9, and/or products containing latex
* have a history of toxic shock syndrome
* have had two or more UTIs in the past year or currently have a suspected or diagnosed UTI or vaginitis by dipstick urinalysis or wet mount, unless treated and proof of cure is documented
* be pregnant, have a suspected pregnancy or desire to become pregnant during the course of the study
* have a history of infertility or conditions which may lead to infertility
* have contraindications to pregnancy (medical condition) or chronic use of class D or X medications
* have been hospitalized for pelvic inflammatory disease without a subsequent intrauterine pregnancy
* have had more than one sexual partner in the past 4 months
* have shared injection drug needles within the past 6 months
* have, or suspected to have, HIV infection
* have been diagnosed with genital herpes simplex virus (HSV), with the first occurrence (initial episode) within the 3 months prior to screening, or have clinical evidence of HSV on exam
* have been diagnosed with any other STDs (including trichomonas) in the 6 months prior to the screening visit
* be lactating or breastfeeding have had a Depo-Provera injection in the 10 months prior to screening
* have a vaginal or cervical abnormality that would interfere with the proper placement and retention of test product and diaphragm

In addition, in order to be eligible to participate in the trial, potential subjects must state that, to her best knowledge, her sexual partner meets the following criteria:

* is not infertile
* has not been treated for Chlamydia trachomatis or N. gonorrhoeae in the past 6 months
* has not been previously diagnosed with, or suspected to have, HIV infection
* has not had more than one sexual partner in the past 4 months
* has not engaged in homosexual intercourse in the past 10 years
* has not shared injection drug needles in the past 10 years
* has no history of allergy or sensitivity to spermicides or products containing N-9
* has no history of allergy or sensitivity to products containing latex

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200
Dates: Start 2004-01; Study Completion 2006-05

PRIMARY OUTCOMES:
Contraceptive efficacy (pregnancy rate) at six months (183 days).